CLINICAL TRIAL: NCT00897481
Title: A Retrospective Case-Control Study of Melanoma Patients Who Have Undergone Sentinel Lymph Node Biopsy
Brief Title: Studying Tumor Tissue Samples From Patients With Melanoma Who Have Undergone Sentinel Lymph Node Biopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leeds Cancer Centre at St. James's University Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CRUK-LCC-06/Q1206/149; CDR0000532943 (Registry Identifier: PDQ (Physician Data Query)); EU-20706
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2008-04

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma; stage IA melanoma; stage IB melanoma; stage IIA melanoma; stage IIB melanoma; stage IIC melanoma; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma
MeSH Terms: conditions — Melanoma | interventions — Gene Expression Profiling; Immunohistochemistry; Sentinel Lymph Node Biopsy

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: mutation analysis
Other: diagnostic laboratory biomarker analysis
Other: immunohistochemistry staining method
Procedure: sentinel lymph node biopsy

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help the study of cancer in the future.

PURPOSE: This laboratory study is looking at tumor tissue samples from patients with melanoma who have undergone sentinel lymph node biopsy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop a predictive model for sentinel lymph node biopsy positivity in patients with melanoma who have undergone sentinel lymph node biopsy.
* Develop a survival model for relapse based on sentinel lymph node biopsy positivity.
* Assess the genetic determinants in primary melanomas that predict a metastatic phenotype and thereby improve understanding of the biology of the metastases in melanoma.

OUTLINE: This is a retrospective, case-controlled, multicenter study. Patients are stratified according to Breslow thickness of the tumor (0.75-1.50 mm vs 1.51- 4 mm vs > 4 mm) and gender.

Archived tumor tissue is analyzed by immunohistochemistry (IHC) for AP2, vascular endothelial growth factor, MMP 2, MCM4, and others, if feasible. Sentinel node biopsies are analyzed by IHC for CD31, LYVE-1, and D2-40 expression. RNA and DNA are also extracted for genetic expression studies and mutation analysis (e.g., BRAF, NRAS, PTEN, CDKN2A).

Patient data related to relapse and recurrence is collected, if available.

Peer reviewed and funded or endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 1,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of cutaneous melanoma

  * Breslow thickness > 0.75 mm
* Has undergone sentinel lymph node biopsy
* No primary melanoma that has not originated in the skin
* No multiple primary melanomas
* Currently under clinical followup OR discharged from follow up within the past 3 months

PATIENT CHARACTERISTICS:

* No other malignancy except for nonmelanoma skin cancer or cervical carcinoma in situ

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Predictive model for sentinel lymph node biopsy positivity
Survival model for relapse
Genetic determinants in primary melanomas that predict a metastatic phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Julia Newton Bishop, MD, Study Chair — Leeds Cancer Centre at St. James's University Hospital
Locations (1):
- Leeds Cancer Centre at St. James's University Hospital, Leeds, England, United Kingdom